CLINICAL TRIAL: NCT06174571
Title: Evaluation of Pregnancy Associated Plasma Protein A (PAPPA) as a Biomarker in Breast Cancer.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Hassan Abdulhady, Assistant Lecturer, Assiut University
Other Study IDs: PAPPA & breast cancer
Record Dates: First submitted 2023-12-02; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: patients diagnosed with breast cancer at different stages of the disease.
- 2: apparently healthy females as a control group.

SUMMARY:
This work aims to:

1. Evaluation of the role of pregnancy associated plasma protein A( PAPPA ) in diagnosis & early detection of breast cancer.
2. Evaluation of the relationship between ( PAPPA ) levels and stages of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* female patients with breast cancer who were diagnosed by histopathological studies and did not receive any treatment.

Exclusion Criteria:

* Patients who received chemotherapy or radiotherapy.
* Patients with known other organ malignancy.

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: female patients with breast cancer at different stages of the disease.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative measurement of pregnancy associated plasma protein A in female patients with breast cancer. | baseline
  Quantitative measurement of pregnancy associated plasma protein A in female patients with breast cancer.